CLINICAL TRIAL: NCT01489878
Title: Impact of Ambulatory Antibiotics Use on Nasal Carriage of Methicillin-resistant Staphylococci in Community Patients : the StaphMRG Study
Brief Title: Antibiotics Use and Carriage of Methicillin-resistant Staphylococci in Community Patients
Acronym: StaphMRG
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081118; 2009-AO1344-53 (Other: french ministry)
Record Dates: First submitted 2011-12-05; First posted 2011-12-12 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Methicillin Resistant Staphylococcus Aureus
Keywords: Coagulase-negative staphylococci; Staphylococcus epidermidis; Staphylococcus aureus; Anti-bacterial agents; Drug resistance, Microbial; Methicillin resistance; Β-lactams; Fluoroquinolones; Macrolides; Synergistin; General practitioners; Antibiotic selection pressure; Ambulatory antibiotherapy; Community patients
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Three samples of nasal flora should be obtained for each included patient: (i) the first one before antibiotic exposure (at inclusion, by the patient's GP) (ii) the second and third ones at the GP's office at the end and 23 to 45 days after the termination of antibiotherapy, respectively.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- β-lactams: amoxicillin-clavulanate or penicillins M
- macrolides
- fluoroquinolones
- synergistins

SUMMARY:
In this prospective, observational, multicentric open study, the investigators will compare the acquisition rates of methicillin-resistant staphylococci (coagulase-negative staphylococci and Staphylococcus aureus) nasal carriage in community patients receiving an ambulatory antibiotic treatment by either a β-lactam (amoxicillin-clavulanate or penicillins M), a macrolide, a synergistin or a fluoroquinolone.

DETAILED DESCRIPTION:
Rationale: Recent spread of community-acquired, methicillin-resistant Staphylococcus aureus (CA-MRSA) represents a major Public Health concern. MR coagulase-negative staphylococci (MR-CoNS) are a likely reservoir of the MR determinant Staphylococcal Cassette Chromosome mec (SCCmec) for S. aureus (SA). Amoxicillin-clavulanic acid, penicillins M, macrolides and synergistin are the most prescribed antistaphylococcal antibiotics in the French community, but their respective impacts on nasal colonization by MR-CoNS and SA have not been investigated in this population.

Primary objective: To compare the acquisition rate of MR-CoNS nasal carriage in community patients treated by β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones at the end of antibiotherapy.

Secondary objectives: (i) To compare the acquisition rate of MR-CoNS nasal carriage in community patients treated by β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones 23 to 45 days after the end of antibiotherapy; (ii) To describe the frequency of co-colonization by SA and MR-CoNS after antibiotic use; (iii) To compare the selection pressure of these 4 classes of antibiotics in term of antibiotic resistances associated to MR in carriage strains of staphylococci (iv) To assess the biodiversity of SCCmec in community-acquired MR-CoNS.

Sudy design and methods: investigators propose to perform a prospective, multicentric study of MR staphylococci carriage in community patients receiving antibiotics prescribed by their general practitioner (GP). Patients older than 18, treated by β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones for a minimal expected duration of 5 days (whatever the indication) and consenting to the study protocol will be eligible for inclusion. Hospitalization within the previous 6 months, antibiotherapy within the previous 2 months, and second line antibiotherapy after inclusion will constitute exclusion criterions. Demographic and medical data will be collected at inclusion. Three samples of nasal flora should be obtained for each included patient: (i) the first one before antibiotic exposure (at inclusion, by the patient's GP) (ii) the second and third ones at the GP's office at the end and 23 to 45 days after the termination of antibiotherapy, respectively. Enrolled patients will participate to the study for 5 to 7 weeks, depending on the duration of antibiotherapy. Samples will be transferred to the Bacteriology unit of the BICHAT-Claude Bernard hospital for MR-CoNS and S. aureus carriages screening, antibiotic susceptibility testing and SCCmec characterization by multiplex PCR.

Number of patients (duration of the study), statistical analysis: Carriage rate of MR-CoNS in the community is 10%-20%. Expected acquisition rates are 20% for patients treated by penicillin M and amoxicilline-clavulanic acid, and less than 5% for patients treated by synergistin. Acquisition rate is not predictable in the macrolides group. To demonstrate a significant difference in acquisition rates (power = 90%, α risk = 5%), 578 patients should definitively be included (141 in each group, including an anticipated 25%-rate of patients lost to follow-up), for a total study duration of 22 months.

Number of participating GP: 48 GP from Paris and its suburb, and affiliated with the Department of General Medicine of BICHAT medical school-Paris 7 University.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age older than 18
* Prescription by a General Practitioner (investigator) of a β-lactam (amoxicillin-clavulanate or penicillins M), a macrolide, a synergistin or a fluoroquinolone for a minimal expected duration of 5 days (whatever the indication)
* Informed consent to the study protocol

NON-INCLUSION CRITERIA:

* Hospitalization within the previous 6 months
* Antibiotherapy within the previous 2 months
* Combination antibiotherapy

EXCLUSION CRITERIA:

* Prescription of a second-line antibiotherapy after inclusion
* Withdrawal of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: community patients receiving antibiotics prescribed by their general practitioner (GP). Patients older than 18, treated by β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistins or fluoroquinolones for a minimal expected duration of 5 days (whatever the indication) Hospitalization within the previous 6 months, antibiotherapy within the previous 2 months, and second line antbiotherapy after inclusion will constitute exclusion criterions.
Sampling Method: Non-Probability Sample
Enrollment: 571 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Short-term impact of ambulatory use of β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones on MR-CoNS nasal carriage in community patients | Between 5 days and 15 days
  assessment of MR-CoNS carriage by nasal swabbing immediately before antibiotic use and within the 3 days following the scheduled end of antibiotherapy - comparison of acquisition rates between the 4 groups (β-lactams, macrolides, synergistin or fluoroquinolones)

SECONDARY OUTCOMES:
Mid-term impact of ambulatory use of β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones on MR-CoNS nasal carriage in community patients | 23 to 45 days after the scheduled end of antibiotherapy (prescribed duration)
  assessment of MR-CoNS carriage by nasal swabbing immediately before antibiotic use and 23 to 45 days after the scheduled end of antibiotherapy - comparison of acquisition rates between the 4 groups
Short-term and mid-term impacts of ambulatory use of β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones on SA and MR-CoNS nasal co-carriage in community patients | within 3 days and 23 to 45 days after the scheduled end of antibiotherapy (prescribed duration)
  assessment of SA and MR-CoNS co-carriage by nasal swabbing immediately before antibiotic use, and within the 3 days and 23 to 45 days after the scheduled end of antibiotherapy - comparison of rates of co-carriage between the 4 groups
Comparison of selection pressure of ambulatory use of β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones in terms of non-β-lactams resistances in MR-CoNS isolates colonizing community patients | within 3 days and 23 to 45 days after the scheduled end of antibiotherapy (prescribed duration
  assessment of non-β-lactams resistances in nasal carriage isolates of MR-CoNS colonizing community patients immediately before antibiotic use, and within the 3 days and 23 to 45 days after the scheduled end of antibiotherapy - comparison of selection pressures between the 4 groups
Short-term and mid-term impacts of ambulatory use of β-lactams (amoxicillin-clavulanate or penicillins M), macrolides, synergistin or fluoroquinolones on the biodiversity (species, SCCmec elements) of MR-CoNS isolates colonizing community patients | within 3 days and 23 to 45 days after the scheduled end of antibiotherapy (prescribed duration)
  assessment of the biodiversity (species, SCCmec elements) of nasal carriage isolates of MR-CoNS colonizing community patients immediately before antibiotic use, and within the 3 days and 23 to 45 days after the scheduled end of antibiotherapy - biodiversity comparison between the 4 groups

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Ruimy, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat-Claude Bernard teaching hospital (AP-HP) and Xavier Bichat medical school (Denis Diderot - Paris 7 university), Paris, France